CLINICAL TRIAL: NCT02989116
Title: Executive Training and Brain in School-Age Children
Brief Title: Executive Training and Brain in Children
Acronym: APEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015-A00383-46; 15-045 (Other: University Hospital, Caen)
Record Dates: First submitted 2016-05-27; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Children; Preterm Birth
Keywords: Learning; Executive functions; Cognitive control; Prefrontal Cortex; Typically developing children; Genotype; Functional Magnetic Resonance Imaging; Structural Magnetic Resonance Imaging; Inhibition; Working Memory; Metacognition; Mindfulness; Preterm children; Developmental Psychology; Developmental cognitive neuroscience; Touch screen tablet; Adaptive training
MeSH Terms: conditions — Premature Birth; Inhibition, Psychological | interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Preterm Inhibition (Experimental): In children born very preterm:
  Inhibition training, Saliva collection, Brain Magnetic Resonance Imaging, Cognitive testing
  Interventions: Behavioral: Inhibition training; Genetic: Saliva collection; Procedure: Brain Magnetic Resonance Imaging; Behavioral: Cognitive testing
- Full-term Inhibition (Experimental): In children born full-term:
  Inhibition training, Saliva collection, Brain Magnetic Resonance Imaging, Cognitive testing
  Interventions: Behavioral: Inhibition training; Genetic: Saliva collection; Procedure: Brain Magnetic Resonance Imaging; Behavioral: Cognitive testing
- Full-term Working memory (Experimental): In children born full-term:
  Working memory training, Saliva collection, Brain Magnetic Resonance Imaging, Cognitive testing
  Interventions: Behavioral: Working memory training; Genetic: Saliva collection; Procedure: Brain Magnetic Resonance Imaging; Behavioral: Cognitive testing
- Full-term Mindfulness (Experimental): In children born full-term:
  Mindfulness training, Saliva collection, Brain Magnetic Resonance Imaging, Cognitive testing
  Interventions: Behavioral: Mindfulness training; Genetic: Saliva collection; Procedure: Brain Magnetic Resonance Imaging; Behavioral: Cognitive testing
- Full-term Active control (Active Comparator): In children born full-term:
  Active control training, Saliva collection, Brain Magnetic Resonance Imaging, Cognitive testing
  Interventions: Behavioral: Active control training; Genetic: Saliva collection; Procedure: Brain Magnetic Resonance Imaging; Behavioral: Cognitive testing

INTERVENTIONS:
Behavioral: Inhibition training — Inhibition training on a tactile tablet for a month (20 sessions of 15 min)
  Arms: Full-term Inhibition; Preterm Inhibition
Behavioral: Working memory training — Working memory training on a tactile tablet for a month (20 sessions of 15 min)
  Arms: Full-term Working memory
Behavioral: Mindfulness training — Mindfulness training on a tactile tablet for a month (20 sessions of 15 min)
  Arms: Full-term Mindfulness
Behavioral: Active control training — Active control training on a tactile tablet for a month (20 sessions of 15 min)
  Arms: Full-term Active control
Genetic: Saliva collection — Collection of a saliva sample for genotyping
Procedure: Brain Magnetic Resonance Imaging — Structural and functional MRI
Behavioral: Cognitive testing — Battery of cognitive and academic tasks on executive functions

SUMMARY:
The purpose of this study is to determine whether a daily executive training to cognitive inhibition, working memory or mindfulness as compared to an active control condition has a near- and far-transfer impact on brain and behavioral measures as collected in children aged 9-10 years, either born preterm or full-term.

ELIGIBILITY:
Inclusion Criteria for all children:

* Male or female
* Aged 9-10 years at inclusion
* French school curriculum (since 1st grade)
* Fully informed through the dedicated booklet
* Both parents gave their written consent
* Normal medical, neurological and brain imaging assessment

Inclusion criterion for non preterm children only:

- Full term pregnancy with no abnormal event (>= 37 weeks of amenorrhea)

Inclusion criterion for preterm children only:

- Delivery before 33 weeks of amenorrhea

Exclusion Criteria for all participants:

* Age over or under 9-10 years old at inclusion
* Monozygotic twins
* Restrictions to a Magnetic Resonance brain imaging exam: claustrophobia, metallic elements (cardiac implants, cochlear implants, metallic elements in the brain or the eyes and being close to the nervous system, metallic prothesis, braces), restless participants.
* Sudden cognitive impairments due to a stroke, head injury associated with loss of consciousness for more than one hour or encephalitis.
* Chronic neurological, psychiatric, infectious or liver condition, endocrine disruption.
* Past or current medical condition: cancer, diabetes, chronic lung condition, cardiac, metabolic, hematological, endocrine or immunological disorder.
* Medication assumed to interfere with brain imaging measures (psychotropics, hypnotics, anxiolytics, neuroleptics, benzodiazepine, steroidal anti-inflammatory, anti-epileptics, painkillers, muscle relaxants).
* Left-sided handedness
* Colour blindness or non-corrected visual disturbances
* Diagnosed developmental disorders
* Diagnosed cerebral palsy
* Diagnosed Fine motor disturbances
* Parents not affiliated to the Social Security
* Parents not able to join at each time of the study

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in brain functional BOLD activity after one month of executive training as assessed by MRI in regions subtending executive functioning. | 3 months: Pretest (t0), immediate Post-test (t0+1 month), deferred post-test (t0+3 months)
  Change in brain activation will be measured with functional magnetic resonance imaging (fMRI) during two different tasks: a Stop Signal task assessing inhibition and a Dot task assessing working memory.
Change in brain cortical structure after one month of executive training as assessed by anatomical MRI in regions subtending executive functioning. | 3 months: Pretest (t0), immediate Post-test (t0+1 month), deferred post-test (t0+3 months)
  Change in brain cortical structure will be measured with anatomical magnetic resonance imaging (aMRI) using four different measures:
  2.a. grey matter volume 2.b. cortical thickness 2.c. cortical surface area 2.d. curvature
Change in cognitive behavioral measures after one month of executive training as assessed by cognitive testing | 3 months: Pretest (t0), immediate Post-test (t0+1 month), deferred post-test (t0+3 months)
  The cognitive testing session includes several tasks assessing executive functioning under different conditions. Will be investigated:
  3.a. Response Time 3.b. Accuracy

SECONDARY OUTCOMES:
Sulcal morphometry measured by anatomical MRI | Pretest (t0)
  Assessing the impact of the early determined sulcal morphometry on behavioral and brain changes associated to a one-month executive training.
Genetic variations measured by Single Nucleotide Polymorphism (SNP) genotyping | Pretest (t0)
  Assessing the impact of the different genotypes on behavioral and brain changes associated to a one-month executive training.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Houdé, Professor, Principal Investigator — University of Paris 5 - Rene Descartes
Locations (1):
- GIP Cyceron, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided